CLINICAL TRIAL: NCT04251416
Title: A Phase II Evaluation of Sacituzumab Govitecan (IMMU-132), an Anti-Trop-2-SN-38 Antibody-drug Conjugate, in Patients With Persistent or Recurrent Endometrial Carcinoma
Brief Title: A Study of Sacituzumab Govitecan (IMMU-132) in Endometrial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000026850
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Govitecan (Experimental): Sacituzumab govitecan will be administered at 10 mg/kg weekly as an infusion for 2 consecutive weeks (2 weekly doses plus 1 week without treatment represents a single 3 week cycle). Treatment can be continued without a rest period in the absence of progression of disease or unacceptable toxicity.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab govitecan will be administered at 10 mg/kg weekly as an infusion for 2 consecutive weeks (2 weekly doses plus 1 week without treatment represents a single 3 week cycle). Treatment can be continued without a rest period in the absence of progression of disease or unacceptable toxicity.
  Other Names: IMMU-132

SUMMARY:
This is a non-randomized Phase 2 study of sacituzumab govitecan (IMMU-132) in subjects with persistent or recurrent endometrial carcinoma.

DETAILED DESCRIPTION:
This is an open-label, Phase 2 study designed to assess the clinical activity of sacituzumab govitecan in subjects with persistent or recurrent endometrial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically confirmed (ie, CAT scan and/or MRI) persistent or recurrent EC of epithelial origin that has progressed after prior platinum based chemotherapy or is refractory to platinum-based chemotherapy.

  * Must have availability of archival tumor tissue FFPE block for TROP-2 testing
  * Note: The presence or absence of TROP-2 overexpression will NOT determine eligibility for study enrollment.
* The diagnosis must be histologically confirmed by a gynecologic pathologist.
* All patients must have measurable disease. Measurable disease is defined as lesions which can be measured by physical examination or by means of medical imaging techniques. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation or plain x-ray, or ≥ 10 mm when measured by spiral CT and/or MRI. Ascites and pleural effusions are not to be considered measurable disease.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST v1.1. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence following completion of radiation therapy.
* After undergoing surgery, patients may be optimally or sub optimally debulked.
* Patients with measurable recurrent disease of any previous substage (I-IV) are eligible to enrollment.
* Patients must have adequate bone marrow function: WBC greater than or equal to 3,000/ul, Platelets greater than or equal to 75,000/ul, Neutrophils greater than or equal to 1500/ul.
* Patients must have adequate renal function: creatinine less than or equal to 2.0 mg/dL.
* Patients must have adequate hepatic function: Bilirubin ≤ 1.5 X laboratory normal. SGOT/SGPT ≤ 3 X laboratory normal or ≤ 5 X laboratory normal if known liver metastases.
* Patients must have an ECOG performance status of 0 or 1.
* Patients must have signed an approved informed consent.
* Patients must be at least 2 weeks beyond prior treatment (chemotherapy, investigational drugs including small molecular inhibitors, endocrine therapy, immunotherapy and/or radiation therapy) or major surgery.
* Patients must be at least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids ≤ 20 mg prednisone or equivalent daily are permitted).
* Patients must have recovered from all acute toxicities to Grade 1 or less from adverse events due to a previously administered agent.

  * Note: Patients with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients with recurrent disease may have received multiple prior chemotherapies for treatment of their endometrial cancer.
* Patients may have received prior immunotherapy therapy alone or in combination with chemotherapy.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the study entry and be practicing an effective form of contraception during the study and until conclusion of 12-week post-treatment evaluation period.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Have an active second malignancy. Note: Patients with a history of malignancy that has been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or subjects with surgically-cured tumors with low risk of recurrence are allowed to enroll.
* Patients with a significant history of cardiac disease within 6 months, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure (NYHA classification III-IV) or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring antiarrhythmia therapy.
* Patients with known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months.
* Patients with any unstable medical issue (including cardiac issues as above, active treatment for symptomatic pulmonary embolism, CVA, renal or hepatic insufficiency, and active infection/sepsis requiring IV antibiotics).
* Have known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤ 20 mg/day of prednisone or its equivalent. All patients with carcinomatous meningitis are excluded regardless of clinical stability.
* Patients who have an uncontrolled seizure disorder, or active neurological disease.
* Have a known history of HIV-1/2 with uncontrolled viral load and on medications that may interfere with SN-38 metabolism.
* Have active HBV or HCV. In subjects with a history of HBV or HCV, subjects with a detectable viral load will be excluded.
* Known hemorrhagic diathesis or active bleeding disorder.
* Patients with Gilbert's disease.
* Patients with active ≥ grade 2 anorexia, nausea or vomiting, diarrhea, and/or signs of intestinal obstruction.
* Prior history of clinically significant bleeding, intestinal obstruction, or GI perforation within 6 months of initiation of study treatment.
* Patients with a history of an anaphylactic reaction to irinotecan or ≥ Grade 3 GI toxicity to prior irinotecan.
* Patients who have previously received topoisomerase I inhibitors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 4 Years
  Objective response rate (complete response and partial response rates) by RECIST1.1 criteria in patients with persistent or recurrent endometrial carcinoma (EC)

SECONDARY OUTCOMES:
Duration of overall survival (OS) | 6 Years
  Overall survival is defined as the duration of time from study entry to death or the date of last contact.
Duration of progression free survival (PFS) | 6 Years
  Progression free survival is defined as the duration of time from study entry to time of progression, death, or is censored at date of last disease assessment
Durable disease control rate (DDCR) | 6 Years
  The percentage of patients who have achieved complete response, partial response, and stable disease
Assess the safety profile of sacituzumab govitecan in endometrial cancer patients (adverse events as assessed by CTCAE v5.0) | 6 Years
  Incidence of treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D. Santin, M.D., Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States